CLINICAL TRIAL: NCT03019263
Title: Nutraceutical Intervention With Berberine, Chlorogenic Acid and Tocotrienols for Menopause-associated Dyslipidemia: a Randomized, Controlled Trial
Brief Title: Berberine, Chlorogenic Acid and Tocotrienols in Menopause-associated Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140012470
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutraceutical (Experimental): Nutritional counseling plus one pill of an active product (Trixy®) containing Berberine, Tocotrienols and Chlorogenic acid
  Interventions: Dietary Supplement: Nutraceutical
- Control (Active Comparator): Nutritional counseling
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Nutraceutical — Nutritional counseling plus one pill of an active product (Trixy®) containing Berberine, Tocotrienols and Chlorogenic acid
  Arms: Nutraceutical
Other: Control — Nutritional counseling
  Arms: Control

SUMMARY:
Menopause is usually associated with an increase in body weight, a change in body composition and fat distribution and a large number of cardio-metabolic changes, such as hypertension, reduction of insulin-sensitivity and dyslipidaemia. The first-line strategy for these complications is the modification of dietary habits and lifestyle in terms of physical activity. Besides, there is also a growing interest in complementary therapies (i.e. nutraceuticals) that can be used alone or in combination to achieve more consistent results. In this context, preliminary evidence supports the potential role of some compounds of vegetal origin such as berberine, chlorogenic acid and tocotrienols. However, in support of their use, the evidence from good quality trials is limited.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol >100 mg/dL
* Written informed consent available

Exclusion Criteria:

* Use of any drug affecting blood lipids
* Hormone replacement therapy
* Adherence to a weigh loss diet in the previous 6 months
* Cancer diagnosis
* Known thyroid, liver, renal or muscle diseases
* Any medical or surgical condition which could lead to an inconstant adhesion to the protocol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 3 months
  LDL cholesterol

SECONDARY OUTCOMES:
Insulin resistance | 3 months
  Homeostatic model assessment (HOMA index)
Total cholesterol | 3 months
  Total cholesterol
HDL cholesterol | 3 months
  HDL cholesterol
Blood glucose | 3 months
  Blood glucose
Serum Insulin | 3 months
  Serum Insulin
Body weight | 3 months
  Body weight
Fat distribution | 3 months
  Waist circumference
Fat Mass | 3 months
  Fat Mass
Menopausal symptoms | 3 months
  Greene Climacteric Scale
Quality of life | 3 months
  36-Item Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided